CLINICAL TRIAL: NCT00820482
Title: A Prospective, Randomized, Controlled Trial Comparing Highly Purified hMG With Recombinant FSH + Recombinant LH in Women Undergoing Intrauterine Insemination: Ovarian Response and Clinical Outcomes.
Brief Title: Comparing Highly Purified hMG With Recombinant FSH + Recombinant LH in Women Undergoing Intrauterine Insemination.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Dr. Elena Labarta, Instituto Valenciano de Infertilidad, Spain
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VLC- EL-0106-307-9
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Ovarian Stimulation Preceding Intrauterine Insemination
MeSH Terms: interventions — Menotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Group A: 75 UI/day of Hp-hMG (Menopur®, Ferring, Copenhaghen, Dinamarca)
  Interventions: Drug: Menopur®, Ferring
- Group B (Experimental): 75UI/day of rFSH (Gonal®, Serono, Ginebra, Suiza) + 75UI/day of rLH (Luveris®, Serono, Ginebra, Suiza)
  Interventions: Drug: rFSH (Gonal®,

INTERVENTIONS:
Drug: Menopur®, Ferring — 75 UI/day of Hp-hMG (Menopur®)
  Arms: Group A
Drug: rFSH (Gonal®, — 75UI/day of rFSH (Gonal®, Serono) + 75UI/day of rLH (Luveris®, Serono)
  Arms: Group B

SUMMARY:
The present study aims to elucidate if the FSH and LH activity contained in hMG preparations is comparable to the recombinant FSH and LH administration in a 1:1 ratio. The mean outcome is the corresponding ovarian response in terms of oestradiol increase during stimulation and number of mature follicles the day of hCG administration. The patients will be included and randomized into two groups and stimulated either by HMG injections started on day 3 at a dose of 75 IU every day and fixed for the first 5 days, and in the second group, rFSH and rLH injections be started on day 3 at a dose of 75 UI/day of rFSH + 75UI/day of rLH. Serum estradiol levels will be measured on stimulation day 1, day 6 and the day of hCG injection. All follicles greater than 14 mm of diameter will be recorded on hCG day Intrauterine insemination is performed during two consecutive days starting the day after the human chorionic gonadotrophin (Ovitrelle) injection. Secondary outcomes are Days of stimulation, Total doses of gonadotrophins administrated, Clinical pregnancy , Ongoing pregnancy and Miscarriage rate, and Cancellation rate.

ELIGIBILITY:
Inclusion Criteria:

* Esterility > 1 year duration
* < 39 years old
* REM > 3 millions/ml
* 1 or 2º IUI cycle

Exclusion criteria:

* Ovarian policystic syndrome
* Severe Endometriosis
* Uterine disease (polyps, myomas, intracavitarios, malformations…)

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The present study aims to elucidate if the FSH and LH activity contained in hMG preparations is comparable to the recombinant FSH and LH administration in proporción 1:1. Mean outcome: - Ovarian response according to the protocol used. | one month

SECONDARY OUTCOMES:
Secondary outcomes: - Days of stimulation - Total doses of gonadotrophins administrated - Clinical pregnancy , ongoing pregnancy and miscarriage rate - Cancellation rate | one cycle

CONTACTS AND LOCATIONS:
Overall Officials: Elena Labarta, MD, Principal Investigator — IVI Valencia
Locations (1):
- IVI Valencia, Valencia, Valencia, Spain